CLINICAL TRIAL: NCT05911269
Title: Determining the Feasibility of Virtual, Tailored, Music-Based Relaxation for Anxiety in Adolescent and Young Adult Cancer Survivors
Brief Title: Feasibility of Virtual, Tailored, Music-Based Relaxation for Anxiety in Adolescent and Young Adult Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.024; HUM00231408 (Other: University of Michigan); R34CA286712 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Timbre Perception

STUDY DESIGN:
Intervention Model Description: Explanatory-Sequential Mixed Methods Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TiMBRe (Experimental): an eight-week, (45 min/week), theory driven, virtually-delivered, tailored music-based relaxation (TiMBRe) intervention to decrease anxiety in AYA cancer survivors with clinically-relevant anxiety.
  Interventions: Other: TiMBRe
- Attention-Control (Active Comparator): Standard of care study staff calls and cancer survivorship resources
  Interventions: Other: Control

INTERVENTIONS:
Other: TiMBRe — 1 & 2 Music Listening
  * Live music played by the music therapist (e.g., guitar, voice) and AYA selected music will be used to facilitate attention to the present moment and provide cues for breathing/relaxation.
    3 & 4 Music Facilitated Breathing
  * The therapist will lead participants in music facilitated breathing exercises using rhythmic features of the music to cue structured breathing for relaxation and self-awareness
    5 & 6 Music Facilitated Progressive Muscle Relaxation for Stress Reduction
  * Using music as a structured auditory cue for tensing and releasing of muscles.
    7 Body Percussion
  * The therapist will lead participants in a hands-on body percussion activity to bring attention to the sound of rhythm, sensation in their hands and body.
    8 Participants Choice
  * will be selected by the participant.
  Arms: TiMBRe
Other: Control — Standard of care study staff calls and cancer survivorship resources
  Arms: Attention-Control

SUMMARY:
Demonstrate the feasibility of conducting an eight-week, (45 min/week), theory driven, virtually-delivered, tailored music-based relaxation (TiMBRe) intervention to decrease anxiety in adolescent and young adult (AYA) cancer survivors with clinically-relevant anxiety.

DETAILED DESCRIPTION:
Initially Sessions 7 and 8 were both body percussion; however, the 04FEB2025 changed this to Session 7 will be body percussion and session 8 will be selected by the participant. This will allow for more tailoring of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 15 - 39 years old
* at least one month post cancer treatment
* report clinically relevant anxiety in the past seven days (PROMIS Anxiety 4a scores ≥ 55)35
* speak/read English.

Exclusion Criteria:

* prognosis less than 3 months
* documentation of significant hearing impairment
* plan to receive surgery, radiation, or chemotherapy for cancer treatment during the study period
* plans in place to begin new psychosocial (i.e., cognitive behavioral therapy14 or mindfulness-based stress reduction15) or pharmacological treatments for anxiety during the study. Although, participants may continue psychosocial or pharmacological treatments for anxiety if the treatments were initiated at least eight weeks prior to study enrollment, the dose has not changed, and they report clinically relevant anxiety in the last week.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of TiMBRe | up to 8 weeks post start of intervention
  mean scores for the Acceptability E-scale Items are ≥ 4/5
Demand of TiMBRe | up to 3 years from start of study
  percent of patients recruited over three years
Adherence to TiMBRe | From enrollment to end of treatment at 8 weeks
  percent of TiMBRe participants to complete the baseline and 8 weeks patient report measures
Practicality of TiMBRe | From enrollment to end of treatment at 8 weeks
  percent of TiMBRe group participants self-report practicing music-based relaxation skills for at least 10 minutes on at least three days per week

SECONDARY OUTCOMES:
Identification of facilitators and barriers to virtual TiMBRe participation | up to 8 weeks post start of intervention
  Interviews will be transcribed by a professional HIPAA compliant transcription agency. We will analyze interview data using inductive content analysis.74 Transcripts will be entered into NVivo Qualitative Data Analysis Software (QSR International, Melbourne, Australia). The study team will read transcripts to derive codes, discuss labels to group codes into categories, and identify major themes and corresponding exemplar quotes. The interviewer will write reflexive memos after each interview and review memos with corresponding audio recordings to discern linkages, gaps, and questions.
Change in Anxiety management | at baseline and eight weeks post initiation of treatment
  determine the preliminary impact of the eight-week virtual TiMBRe intervention, relative to the control, on improving anxiety (PROMIS Anxiety 4a, 40.3 - 81.6; higher scores = worse anxiety) utilizing data collected at baseline, four weeks, and eight weeks. Reporting the change from baseline to eight weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No